CLINICAL TRIAL: NCT00324532
Title: An Open Label, Non Comparative, Prospective Pilot Study, to Assess the Efficacy and Safety of the Probiotic E. Coli Strain M17 on Patients With GERD
Brief Title: to Assess the Efficacy and Safety of the Probiotic E. Coli Strain M17 on Patients With GERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioBalance Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB 07 2005
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2006-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Drug: ProBactrix

SUMMARY:
The study is an Open Label, Prospective, Non Comparative, Pilot, clinical trial design. Patients with inadequate relief in GI symptoms associated with GERD despite PPI treatment will be screened and those who meet the inclusion and exclusion criteria will perform a glucose breath test for bacterial overgrowth . Each patient will then complete a questionnaire to record their GERD related symptoms. Each patient will then receive a daily intake of 30 mL two times daily, 30 minutes before meals for a period of 4 weeks. During the course of the trial, they will have 4 visits with the study physician to assess treatment compliance and occurrence of adverse events, and will complete periodic daily diaries to record compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between ≥18 and ≤80, males and females.
2. Patient administered PPI therapy for GERD.
3. Patient suffers from any GI symptoms including GERD symptoms despite PPI therapy for at least 60 days
4. Patient with positive or negative glucose breath test for bacterial overgrowth unless they are not able to do this secondary to diabetes. Diabetics will have a lactulose breath test
5. Able to give informed consent
6. Candidate will be available for the next 4 weeks

Exclusion Criteria:

1. Pregnant, breast-feeding, or not using approved methods of contraception (if of childbearing potential) 2. Unstable medical disorder 3. Patient has had E. coli strain M17 administered in the past month 4. History of major psychiatric disorder or substance abuse within the previous 2 years, including psychiatric illnesses requiring medication that may cause doubt in the validity of the signed Informed Consent form 5. Existing illness or medical condition that will prevent the patient from participating in the study (such as severe heart disease, insulin dependent diabetes, hyperactive thyroid gland, HIV positive, etc.) 6. Participation in another clinical study during the past four weeks. 7. Any use of a probiotic supplement within 30 days of the screening period (with the exception of standard food yogurt products) 8. Any use of antibiotics within 30 days of the screening/enrollment period (however, candidate may wait to initiate screening exam until 30 days have lapsed since antibiotic course was completed)

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
improvement in one or more GI symptoms (heartburn, regurgitation, bloating, epigastric pain, abdominal pain and general well being).

SECONDARY OUTCOMES:
symptomatic response comparison between patients with a positive versus negative breath test for bacterial overgrowth
negative breath test for bacterial overgrowth in the patients with positive breath test at entry
safety

CONTACTS AND LOCATIONS:
Overall Officials: Braverman, Principal Investigator — Shaarei Zedek Medical Center
Locations (1):
- Shaarei Zedek Medical Center, Jerusalem, Israel